CLINICAL TRIAL: NCT04700592
Title: A Comparison of Gabapentin and Ketamine in Acute and Chronic Pain After Inguinal Hernia Repair: a Prospective Randomized Study
Brief Title: A Comparison of Gabapentin and Ketamine in Acute and Chronic Pain After Inguinal Hernia Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Tunis El Manar (Other)
Responsible Party: Principal Investigator, Mechaal Benali, Professor, University Tunis El Manar
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UTEM GABA
Record Dates: First submitted 2021-01-02; First posted 2021-01-08 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-05

CONDITIONS: Chronic Pain Following Surgical Procedure for Cancer
Keywords: post operative chronic pain; gabapentin; ketamin; Inguinal Hernia Repair
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gabapentin group (Experimental): group which receives 600 mg of Gabapentin (two tablets) one hour prior to surgery
  Interventions: Other: Gabapentin versus Ketamine
- ketamine group (Experimental): group which receives an injection of ketamine at a dosage of 0.15 mg/Kg before surgery incision
  Interventions: Other: Gabapentin versus Ketamine

INTERVENTIONS:
Other: Gabapentin versus Ketamine — A Comparison of Gabapentin and Ketamine in Acute and Chronic Pain
  Other Names: acute and Chronic Pain

SUMMARY:
Patients were randomized into two groups: Group Gabapentine ( G group) received 600 mg of Gabapentin (two tablets) two hours prior to surgery and saline solution before induction of spinal anesthesia and group Ketamine ( K group) received two placebo tablets and an injection of ketamine at a dosage of 0.15 mg/Kg before induction of spinal anesthesia.. During the surgery, blood pressure and heart rate were monitored. Postoperative analgesia was provided by a PCA morphine. Acute postoperative pain was assessed by a visual analog scale. The incidence of postoperative neuropathic pain was detected by the DN4 questionnaire after one and three months of surgery.

DETAILED DESCRIPTION:
the investigators includes patients aged at least 18 classified as ASA I and II. Patients with significant cardiovascular or central nervous system disease, as well as those with renal or liver failure and those who could not operate the PCA device were not eligible for our study.

Exclusion criteria were patients that had incidents during the surgery such as: an allergic reaction, local anesthetic systemic toxicity or a surgical incident.

Patients were randomized into two groups: Group Gabapentine ( G group) received 600 mg of Gabapentin (two tablets) two hours prior to surgery and saline solution before induction of spinal anesthesia and group Ketamine ( K group) received two placebo tablets and an injection of ketamine at a dosage of 0.15 mg/Kg before induction of spinal anesthesia.

Upon arrival in the operating room, patients were monitored using mean blood pressure, heart rate and peripheral oxygen saturation monitors.

The surgery was performed under spinal anesthesia. Each patient received 10 mg of hyperbaric bupivacaine mixed with 5 µ of sufentanil.

Immediately after the intervention, the patients were transferred to the post anesthesia care unit (PACU) where analgesia was arranged through morphine titration.

After the motor block is lifted, patients were transferred to surgery department where they were connected to a PCA device that provided 1 mg IV bolus injection of morphine at a lockout interval of 7 minutes and with a maximum four-hour limit of 0.5 mg/Kg.

During the hospital stay, acute post-operative pain assessed through the visual analog scale (VAS) at rest and at motion, every 15 minutes in the PACU and then at H2, H6, H12 and H24 postoperative.

The morphine consumption was noted as well as its first demand. Sedation was assessed using the Ramsay score. The occurrence of adverse effects such as nausea and vomiting, dizziness, diarrhea, hallucination and pruritus was also noted.

The first night sleep quality was evaluated through the Spiegel score. After hospital discharge, patients were contacted at one month and three months. The incidence of post-operative neuropathic pain was detected by the DN4 questionnaire. The effect the pain had on their daily activities was also judged.

Statistical analysis:

According to available data (30% occurrence of post-operative chronic pain after inguinal hernia repair (2)), to decrease by 25% this number with a power of 80%, 28 patients were needed in each group.

Statistical analysis was performed with SPSS in its 20 version. Results were expressed as mean, standard variation or median. χ2 test, fisher's exact test and Mann-Whitney test were performed. A P value of < 0.05 was considered as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* ASA I and II
* Inguinal Hernia Repair in non emergent conditions

Exclusion Criteria:

* Patients with significant cardiovascular central nervous system disease, renal or liver failure could not operate the PCA device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-10-02 (Actual); Primary Completion 2021-02-02 (Actual); Study Completion 2021-02-02 (Actual)

PRIMARY OUTCOMES:
postoperative neuropathic pain | three months of surgery
  the DN4 questionnaire

SECONDARY OUTCOMES:
acute pain postoperative | At twenty-four hour postoperative
  the visual analogue scales (VAS) at rest and at motion
Consumption of morphine | At 24 hour postoperative
  measuring consumption by PCA (PATIENT CONTROLLED ANALGESIA)

CONTACTS AND LOCATIONS:
Overall Officials: mechaal benali, PROFESSOR, Principal Investigator — university manar Tunis tunisia
Locations (1):
- Mechaal Benali, Nabeul, Tunisia

IPD SHARING:
Plan to Share IPD: No